| Life-Skills Training Program: Its effect on Self-efficacy among Patients with Substance Use<br>Disorders | | | |
|---|---|---|---|
| | L. I. Chille The initial | D 14 | C-16 -6C |
| Official title of the study: Life-Skills Training Program: Its effect on Self-efficacy among Patients with Substance Use Disorders | | | |
| NCT number: Pending | | | |
| Date of the document: 1/4/2023 | | | |
| | | 4 | 4 (2022 |
| NCT number: | pending | document date: 1/4 | 4/2023 |

Ministry of Health &Population General Secretariat of Mental Heal and Addiction Treatment



# **Informed Consent for Participation in Scientific Research**

Presented only to potential participants in the study

Those who agree to participate:

## 1- Study Title:

Life-Skills Training Program: Its effect on Self-efficacy among

### **Patients with Substance Use Disorders**

# 2- Purpose of the Study:

This study aimed to evaluate the effect of life-skills training program on self-efficacy among patients with substance use disorders

### 3- Data Protection:

Your name will not be used; instead, a code will represent you to ensure your privacy is maintained in all results.

### 4- New Information:

You will be informed of any new information related to the study as it becomes available.

### **5- Ethics Committee:**

This study has been approved by the General Research Ethics Committee at the Faculty of Pharmacy, Ain Shams University, which ensures that all conditions are met to protect your safety and rights.

# **Contact for Emergencies or Questions:**

Researcher: Abdelmouttelb Abdelkawy

Workplace: faculty of Nursing- Ain Shams University

**Phone**: +201066915835

**Email:** abdelmouttelb@nursing.asu.edu.eg

NCT number: pending document date: 1/4/2023

# Life-Skills Training Program: Its effect on Self-efficacy among Patients with Substance Use Disorders

If you have any questions at any time, you may contact the above or send inquiries via email.

Please take sufficient time to review this information sheet and feel free to ask any additional questions before signing this document.

Your signature will confirm your agreement to participate after understanding all the information.

### **Possible Benefits of the Study:**

Acquiring and learning new skills enables me to handle daily vigilance and protect myself from relapses, as well as adapt to various stresses. I fully understand that I have the right to refuse participation or withdraw from study at any time or at any stage without giving a reason and without any negative consequences.

I understand that I may also refuse to provide any information requested without giving reasons and without any penalty.

# **Participant's Consent:**

- The research study has been clearly explained to me.
- I have received a copy of the information sheet.
- All my rights have been fully explained to me.
- I have signed a copy of the consent form to keep.

I voluntarily agree to participate in the study titled Life-Skills Training

# Program: Its effect on Self-efficacy among Patients with Substance

### **Use Disorders**

I understand that the data and information collected on my behalf will be stored and processed in accordance with personal data protection laws. I acknowledge that the research team bears full responsibility for my rights and safety during the study.

I understand that participation is voluntary and that I may withdraw at any time without legal penalty.

I understand that aggregated data will be used without any personal identifiers to ensure confidentiality.

| Participant's Name: _ | | | |
|-----------------------|---------|----------------|----------|
| NCT number: | pending | document date: | 1/4/2023 |

# Life-Skills Training Program: Its effect on Self-efficacy among Patients with Substance Use Disorders Participant's Signature: Date: \_\_\_\_/ \_\_\_\_ / 20\_\_\_\_ Researcher's Name: Position/Title: Researcher's Signature: \_\_\_\_\_ Date: \_\_\_\_/ \_\_\_\_ / 20\_\_\_\_

NCT number: pending document date: 1/4/2023